CLINICAL TRIAL: NCT04329325
Title: Phase II Study of Blinatumomab and Concurrent Oral Tyrosine Kinase Inhibitor Therapy as Consolidation and Maintenance Therapy for Patients With Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia Following Chemotherapy-Sparing Induction
Brief Title: Blinatumomab and Tyrosine Kinase Inhibitor Therapy in People With Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-343
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia; Philadelphia Chromosome-Positive
Keywords: Blinatumomab; Concurrent Oral Tyrosine Kinase Inhibitor; Chemotherapy-Sparing Induction; 19-343
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; Dasatinib; Dexamethasone; Methotrexate

STUDY DESIGN:
Intervention Model Description: This study is an open-label single arm phase II study with a Simon's minimax two-stage for the treatment of adults with newly diagnosed Ph+ ALL.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab & Concurrent Oral Tyrosine Kinase Inhibitor (TKI) (Experimental): Patients may receive steroids and hydroxyurea pre-study entry and receive a 7-day steroid prephase before starting TKI therapy. Planned initial TKI is dasatinib 140 mg daily; dasatinib dose may be reduced or TKI may be changed to a different agent under certain conditions. Induction consists of continuous TKI + 24 days of dexamethasone, followed by taper of dexamethasone, with bone marrow aspirate/biopsy (BMA) and CNS prophylaxis at days 22 and 43. Patients achieving morphologic complete response post-induction proceed to consolidation with up to 3 cycles of blinatumomab (28-day cycles, 14 days between cycles) + TKI, with BMA and CNS prophylaxis between cycles. Patients achieving complete molecular response may proceed to maintenance with up to 4 more cycles of blinatumomab (28-day cycles with 28 days between cycles) + TKI, with CNS prophylaxis between cycles and BMA after cycles 5 and 7. Patients can come off study to undergo allogeneic hematopoietic cell transplantation at any time.
  Interventions: Biological: Blinatumomab; Drug: dasatinib; Drug: dexamethasone; Drug: methotrexate

INTERVENTIONS:
Biological: Blinatumomab — Please see detailed summary.
Drug: dasatinib — Please see detailed summary.
Drug: dexamethasone — Please see detailed summary.
Drug: methotrexate — Please see detailed summary.

SUMMARY:
The purpose of this study is to test whether blinatumomab in combination with TKI therapy (such as dasatinib) is an effective treatment for people with Ph+ ALL. Researchers want to improve the response to standard-of-care treatment of corticosteroids + TKI therapy by adding the study drug, blinatumomab.

DETAILED DESCRIPTION:
PRE-PHASE: Patients may receive corticosteroids and/or hydroxyurea at the discretion of the treating physician prior to beginning induction therapy. A seven-day corticosteroid pre-phase, which can include days of corticosteroid receipt prior to protocol registration, will precede initiation of TKI therapy on day 1. Corticosteroid dose and schedule are at the discretion of the investigator during the pre-phase, with dosing caps of prednisone 120 mg/day, dexamethasone 24 mg/day, or biologic equivalents thereof. In the event the treating investigator feels delaying induction therapy (TKI + dexamethasone) would be unsafe (e.g. ALL progressing despite corticosteroids), the patient may proceed to day 1 (begin TKI + dexamethasone) before completion of 7-day pre-phase if investigator feels delay would be unsafe.

INDUCTION THERAPY: Induction therapy consists of dexamethasone in combination with TKI. TKI therapy will generally begin with dasatinib 140 mg daily (dose changes or transition to alternative TKI permitted subject to the provisions in the protocol). Patients will receive dexamethasone 10 mg/m2/day (up to 24 mg /day) in single or divided doses, days 1-24. Dexamethasone will be tapered days 25-32 (±3 days for start and end of taper); the TKI will be continued during and following the dexamethasone taper. Recommended CNS prophylaxis consists of intrathecal (IT) or intra-Ommaya (IO) methotrexate 12 mg day 22 and day 43 (±7 days); of note, methotrexate 12 mg is recommended though agent/dosing left to discretion of investigator. Hydrocortisone IT may be given along with methotrexate at the discretion of the investigator. Bone marrow evaluations will be performed on days 22 (±3 days) and day 43 (±3 days) and will include minimal residual disease (MRD) assessment by BCR-ABL1 transcript studies and flow cytometry. Under certain circumstances, the induction period may be extended for up to 21 days with bone marrow studies repeated at that time.

CONSOLIDATION THERAPY: Patients in complete response (CR) or CR with incomplete hematologic recovery (CRi) following remission induction, with or without MRD, proceed to consolidation therapy, defined as day 1 of cycle 1 of blinatumomab, within 21 days of day 43 or the date of BMA establishing CR/CRi, whichever is later. TKI will be administered continuously. Patients will begin Blinatumomab 28 mcg/daily IVCI for patients ≥45 kg; patients <45 kg will be treated at a dose of 15 mcg/m2/day, capped at a dose of 28 mcg/day, given for a 28-day cycle, with dose adjustments further subject to the provisions outlined in the protocol. Inpatient admission is recommended for at least days 1-3 of cycle 1 of blinatumomab (≥72 hours from start of infusion). Following each 28-day infusion of blinatumomab, a mandatory period of 14 days off blinatumomab will follow during which bone marrow evaluation will be performed with MRD assessment and CNS prophylaxis will be administered. The consolidation period will consist of 3 cycles of blinatumomab given as such. Patients may come off therapy at any point to undergo allogeneic hematopoietic cell transplantation (alloHCT).

MAINTENANCE THERAPY: Patients in complete molecular response (as defined within the protocol) following blinatumomab cycle 3 and not proceeding immediately to alloHCT may proceed to maintenance therapy, defined as day 1 of cycle 4 of blinatumomab, within 28 days of completion of blinatumomab infusion in cycle 3. TKI will be administered continuously. Blinatumomab will be given for up to 4 additional 28-day cycles (cycles 4-7) with a mandatory period of 28 days (±7 days) off blinatumomab between cycles, during which CNS prophylaxis will be administered. Bone marrow evaluation with MRD assessment will be performed after cycles 5 and 7 of blinatumomab.

FOLLOW-UP: TKI maintenance is recommended but not required. Further post-remission therapy, if any, at the discretion of the treating physician. Following completion of all required study treatments and assessments, patients enrolled will be followed for long-term survival and relapse outcomes as outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Age ≥ 18 years of age
* Direct bilirubin ≤2x upper limit of normal (ULN), AST and ALT ≤10x upper limit of normal (ULN). Higher bilirubin and AST/ALT levels are acceptable if thought related to Ph+ ALL.
* Histology confirmed by enrolling institution Confirmed diagnosis of acute lymphoblastic leukemia (ALL) by morphology, immunohistochemistry, and/or multiparameter flow cytometry, with confirmation of Philadelphia chromosome positivity (Ph+) by cytogenetic studies (karyotype/FISH), molecular studies (BCRABL1 fusion transcripts), or targeted RNA sequencing
* No prior therapy for ALL beyond corticosteroids, hydroxyurea, or prophylactic intrathecal/intra-Ommaya chemotherapy Acceptable end-organ function (i.e. not meeting exclusion criteria below)
* Amenable to practicing an effective method of birth control during treatment and for at least 3 months following treatment on study
* ECOG performance status 0-2

Exclusion Criteria:

* Philadelphia chromosome-negative ALL
* Mature B-cell ALL (e.g. Burkitt leukemia/lymphoma)
* Active extramedullary disease at time of study entry, including known CNS-3 disease (≥5 WBC/microliter and positive cytology or flow cytometry). Note: LP and/or CNS imaging prior to treatment initiation is not required, but if the patient is found to have active CNS-3 disease (by LP) or evidence of CNS involvement on imaging in the course of evaluation of clinical findings, enrollment is not permissible.
* Presence of known ABL kinase mutations conferring resistance to dasatinib at time of study entry, including T315I mutation. Note: ABL mutation testing prior to treatment initiation is neither recommended nor required, but if results of such mutation testing are known, enrollment of a patient with known ABL kinase mutations conferring dasatinib resistance is not permissible.
* Unable to tolerate oral medication.
* Creatinine >1.5x upper limit of normal and estimated GFR <30 mL/min (based on 24-hour urine collection to determine creatine clearance or CKD-EPI equation) NOTE: Meeting EITHER the blood creatinine level standard OR the estimated GFR standard (based on 24 hour urine collection OR CKD-EPI equation) is required for eligibility. Subjects are excluded only if BOTH criteria are not met.
* Heart disease meeting one or more of the following criteria:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction <6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia
  * History of cardiomyopathy with left ventricular ejection fraction ≤20%
  * Pre-treatment Fredericia-adjusted QTc (QTcF) of >500 msec, unless the patient is thought to be an acceptable candidate for dasatinib after consultation with a cardiologist (including, but not limited to situations in which QTcF is thought not representative of true length of repolarization due to pre-existing bundle branch block or ventricular pacing)
* Patients with active hepatitis B infection (as manifest by either detectable hepatitis B virus DNA by PCR and/or positivity for hepatitis B surface antigen) are ineligible
* Patients with active hepatitis C infection (as manifest by detectable hepatitis C virus RNA by PCR) are ineligible. Patients with detectable antibodies to hepatitis C virus will be screened by PCR for evidence of active infection.
* Patients with HIV infection are ineligible, unless on antiretroviral therapy with undetectable HIV RNA by PCR (using an assay with sensitivity to detect levels of ≥50 copies/mL) and otherwise eligible in the determination of the investigator.
* Ongoing need for systemic T-cell suppressive therapy (e.g. corticosteroids, tacrolimus, cyclosporine for active autoimmune disease or prior solid organ transplantation)
* Concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of skin
* Uncontrolled systemic fungal, bacterial, viral or other infection
* History or presence of uncontrolled or clinically significant neurological disorders such as generalized seizure disorder or severe brain injury
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of evaluable patients achieving complete molecular response | 7 months
  (MRD negativity by flow cytometry and quantitative PCR of BCR-ABL transcripts) at any time during TKI + corticosteroid induction or consolidation with up to 3 cycles of blinatumomab in combination with TKI.

SECONDARY OUTCOMES:
Frequency, severity, and co-occurrence of treatment-related grade 3-4 toxicities | 13 months
  assessed by NCI CTCAE v5.0 and rates of blinatumomab discontinuation due to toxicity among all patients beginning the consolidation portion of the study on dasatinib. The window for toxicity evaluation for this objective extends from the beginning of consolidation of the study until completion of maintenance or removal from study, whichever is sooner."
Proportion of evaluable patients with CMR or molecular MRD positivity with MRD negativity by flow cytometry at any time during induction or consolidation. | 7 months
Duration of CMR among patients achieving MRD negativity after TKI + corticosteroid induction, followed by 1-3 cycles of blinatumomab in combination with an oral TKI. | 2 years
Cumulative incidence of morphologic and molecular relapse following consolidative therapy with blinatumomab in combination with an oral TKI | 2 years
Event-free survival following consolidative therapy with blinatumomab in combination with an oral TKI. | 2 years
Overall survival following consolidative therapy with blinatumomab in combination with an oral TKI. | 2 years
The proportion of patients first achieving CMR at any point during induction and proportion of patients not achieving CMR in Part 1 who subsequently achieved CMR at any point during consolidation. | 7 months

OTHER OUTCOMES:
Frequency, type, and co-occurrence of ABL kinase mutations | 2 years
  As assessed by sequencing of the ABL kinase gene in bone marrow or peripheral blood, observed in patients experiencing progression of B-ALL following consolidative therapy with blinatumomab in combination with an oral TKI.
Frequency, type, and co-occurrence of new somatic mutations | 2 years
  As assessed by next-generation sequencing of bone marrow or peripheral blood, in patients experiencing progression of B-ALL following consolidative therapy with blinatumomab in combination with an oral TKI.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Geyer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm